CLINICAL TRIAL: NCT00854152
Title: An Open-label, Phase I, Dose-Escalation Study Evaluating the Safety, Tolerability, and Maximally Tolerated Dose of GDC-0980 Administered Once Daily in Patients With Refractory Solid Tumors and Non-Hodgkin's Lymphoma
Brief Title: A Study Evaluating GDC-0980 Administered Once Daily in Patients With Refractory Solid Tumors or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIM4604g; MP00880 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma, Solid Cancers
Keywords: NHL; Tumors; Carcinogenic Tumors
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms | interventions — 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GDC-0980

INTERVENTIONS:
Drug: GDC-0980 — Escalating repeating dose

SUMMARY:
This is an open-label, multicenter, Phase I study to evaluate the safety, tolerability, and pharmacokinetics of escalating oral doses of GDC-0980 administered to patients with incurable, locally advanced or metastatic solid malignancy or NHL that has progressed or failed to respond to at least one prior regimen or for which there is no standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, incurable, locally advanced or metastatic solid malignancies, or NHL without leukemic phase, that has progressed despite standard of care therapy or for which there is no standard therapy of proven clinical benefit
* ECOG performance status of 0 or 1 at screening
* Evaluable or measurable disease per RECIST and/or the following: prostate cancer patients with non-measurable disease are eligible if they have two rising prostate-specific antigen (PSA) levels that meet the PSA Working Group criteria for progression prior to initiation of study treatment; ovarian cancer patients with non-measurable disease are eligible if they have two rising CA-125 levels greater than the ULN >= 2 weeks apart prior to initiation of study treatment.
* Life expectancy >=12 weeks
* Adequate hematologic and organ function within 14 days before initiation of GDC-0980
* Documented willingness to use an effective means of contraception for both men and women while participating in the study

Exclusion Criteria:

* Leptomeningeal disease as the only manifestation of the current malignancy
* History of Type 1 or 2 diabetes mellitus requiring regular medication
* Grade >= 2 hypercholesterolemia or hypertriglyceridemia
* Ejection fraction that is <50% or below the LLN (whichever is higher), as determined by echocardiogram or MUGA scan
* DLCO < 50% of predicted value corrected for hemoglobin and alveolar volume prior to initiation of GDC-0980
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Known untreated malignancies of the brain or spinal cord, or treated brain metastases that are not radiographically stable for >= 3 months
* Active congestive heart failure or ventricular arrhythmia requiring medication
* Active infection requiring IV antibiotics
* Requirement for any daily supplemental oxygen
* Uncontrolled hypomagnesemia
* Hypercalcemia requiring continued use of bisphosphonate therapy
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Uncontrolled ascites requiring frequent paracentesis
* Known HIV infection
* Any other diseases, active or controlled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug
* Significant traumatic injury within 4 weeks of Day 1
* Major surgical procedure within 4 weeks prior to initiation of GDC-0980
* For all patients participating in Stage 2: Prior treatment with any PI3K inhibitor, mTOR inhibitor or dual PI3K/mTOR inhibitor. For HNSCC patients, this restriction applies only to any PI3K inhibitor, mTOR inhibitor, or dual PI3K/mTOR inhibitor used in the palliative setting.
* Treatment with chemotherapy, hormonal therapy (except hormone replacement therapy, oral contraceptives, or GnRH agonists or antagonists for prostate cancer), immunotherapy, biologic therapy, radiation therapy (except palliative radiation to bony metastases), or herbal therapy as cancer therapy within 3 weeks prior to initiation of GDC-0980
* Palliative radiation to bony metastases within 2 weeks prior to initiation of GDC-0980
* Need for chronic corticosteroid therapy of >= 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressant
* Treatment with an investigational agent within 4 weeks prior to initiation of GDC-0980
* Unresolved toxicity from prior therapy except for alopecia and Grade 1 peripheral neuropathy
* Pregnancy or lactation
* For patients participating in DCE-MRI assessments, any contraindication to MRI examination
* For patients with advanced solid tumors or NHL participating in the PPI-effect assessment: Known hypersensitivity to rabeprazole, substituted benzimidazoles, or to any component of the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | Length of study
Occurrence of dose-limiting toxicities | Length of study
PK parameters after doses of GDC-0980 | Length of study
Occurrence of Grade 3 and 4 abnormalities in safety-related laboratory parameters and associated dose of GDC-0980 | Length of study

SECONDARY OUTCOMES:
Best overall response, duration of objective response, and progression-free survival for patients with measurable disease | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Mika Derynck, M.D., Study Director — Genentech, Inc.
Locations (5):
- United States (4):
  - Chicago, Illinois
  - Boston, Massachusetts
  - New York, New York
  - Nashville, Tennessee
- Sutton, United Kingdom

REFERENCES:
- [Derived] Moein A, Jin JY, Wright MR, Alicke B, Wong H. Retrospective Assessment of Translational Pharmacokinetic-Pharmacodynamic Modeling Performance: A Case Study with Apitolisib, a Dual PI3K/mTOR Inhibitor. Drugs R D. 2024 Jun;24(2):155-167. doi: 10.1007/s40268-024-00459-5. Epub 2024 May 3. PMID 38700808